CLINICAL TRIAL: NCT04539561
Title: Evaluation of the Efficacy and Safety of PiQo4 for the Treatment of Hand Pigmentation Using 1064nm PSL and 532nm PSL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Focus Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Focus-PiQo4 Pigmentation-19-02
Record Dates: First submitted 2020-03-10; First posted 2020-09-07 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-03

CONDITIONS: Pigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pigmentation (Experimental): Treatment of Hand Pigmentation Using PiQo4 Laser System
  Interventions: Device: PiQo4 Laser System

INTERVENTIONS:
Device: PiQo4 Laser System — PiQo4 Laser System for treatment of hand pigmentation

SUMMARY:
A total of 20 healthy subjects at a single site, aged 21-70 years old with congenital or acquired challenging/resistant, age/sun-related flat and benign hand pigmentation who wish to improve their skin appearance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Female/Male.
* Age= 21-70 (Adults).
* Fitzpatrick skin phototype = I-V
* Congenital or acquired benign pigmentation on hands.
* Presence of at least three (3) lesions with similar pigmentation intensity in the treatment area in diameters larger than 2 mm.
* Able to read, understand and provide written Informed Consent.
* Able and willing to comply with the treatment/follow-up schedule and requirements.
* Women of child-bearing potential are required to use a reliable method of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, NuvaRing, partner with vasectomy, Implanon or other FDA-approved devices, or abstinence) during the course of the study.

Exclusion Criteria:

* History of post inflammatory pigmentary disorders, particularly a tendency for hyper- or hypo-pigmentation.
* Tanning (artificial or natural) 1 month prior first treatment and during the entire study duration including follow-up.
* Excessive underlying vascular conditions (e.g. dense network of capillaries).
* Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 3 months after completion of breastfeeding.
* Prior skin laser, light or other energy device treatment in treated area within 6 months of initial treatment or during the course of the study.
* Prior ablative resurfacing procedure in treated area with laser or other devices within 12 months of initial treatment or during the course of the study.
* Prior treatment with medium-depth or deeper, chemical peels or dermabrasion in treated area within 3 months of initial treatment or during the course of the study.
* Any other surgery in treated area within 9 months of initial treatment or during the course of the study.
* Hypersensitive to light exposure or the use of photosensitive medication for which light exposure is contraindicated.
* Multiple dysplastic nevi or suspicious pigmentation in area to be treated.
* Presence of underlying tattoo in the treatment area.
* Significant concurrent illness (e.g. uncontrolled diabetes) or any disease state that in the opinion of the Investigator would interfere with the treatment or healing process.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Hands pigmentation change assessed by investigator | 1 month follow up
  Hands pigmentation change assessed by investigator at the 1 month follow up using the 5-point Pigment Improvement Score where score of between 0 and 4 will be assigned (0- No improvement in pigmentation, 1- Trace to mild improvement of some lesions, 2- Moderate response: some lesions lighter, 3- Good response: most lesions much lighter and 4- Excellent response- Most or all lesions much lighter or gone.

CONTACTS AND LOCATIONS:
Locations (1):
- "Sk;N" Clinic, London, United Kingdom